

## STATISTICAL ANALYSIS PLAN

Title: A Pilot Study: A Comparison of Liposomal Bupivacaine ("Exparel<sup>TM</sup>") to Bupivacaine HCl in Tranversus Abdominis Planus ("TAP") Block for Abdominal Gynecologic Surgery

Sponsor: Mark Shahin, MD,

Abington Memorial Hospital, 1 Widener Hanjani Institute for Gynecologic Oncology

215-885-0220

Principal Investigator: Heidi Ching, MD

Abington Memorial Hospital

1200 Old York Road Price MOB Suite 109

215-481-4211 518-813-0526

Statistical analysis was performed by the department statistician in order to calculate the sample size necessary to achieve a statistically significant decrease by 0.5 days in length of stay based on the department's average length of stay for open abdominal surgery (3 days). N was calculated to be 128, 64 in each arm. Microsoft Excel program was then used to create a randomization for either control or intervention for a total of 150 patients to anticipate 15% dropout rate.